CLINICAL TRIAL: NCT01026558
Title: Open-Label, Single Dose, Parallel Group Pharmacokinetic Study of Ceftobiprole in Morbidly Obese and Non-Obese Patients
Brief Title: A Study Evaluating the Pharmacokinetics of Ceftobiprole When Taken by Obese Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CR014185; CSI-1008 (Other: Basilea (Internal Reference))
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2012-08

CONDITIONS: Obesity; Staphylococcal Skin Infections; Streptococcal Infections
Keywords: Obesity, Ceftobiprole; Skin Infections; Staphylococcal Skin Infections; Bacterial Skin Infections; Streptococcal Infection
MeSH Terms: conditions — Obesity; Staphylococcal Skin Infections; Streptococcal Infections; Cellulitis | interventions — ceftobiprole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ceftobiprole (not morbidly obese subjects) (Active Comparator): Ceftobiprole 500 mg single-dose over 2 hours.
  Interventions: Drug: Ceftobiprole
- Ceftobiprole (morbidly obese subjects) (Experimental): Ceftobiprole 500 mg single-dose over 2 hours.
  Interventions: Drug: Ceftobiprole

INTERVENTIONS:
Drug: Ceftobiprole — Ceftobiprole, 500 mg as single iv infusion over 2 hours

SUMMARY:
The primary objective of this study is to compare the pharmacokinetics (how drugs are absorbed in the body, how they are distributed within the body and how they are removed from the body over time) of ceftobiprole in morbidly obese patients and non-obese patients. The secondary objectives are to assess the pharmacodynamics (the study of the action or effects a drug has on the body) and to assess safety and tolerability of ceftobiprole in order to support dosing recommendations in the morbidly obese population.

DETAILED DESCRIPTION:
This is an open-label (all people involved know the identity of the intervention), parallel-group, Phase 1 study in morbidly obese and non-obese men and women. A total of 25 patients (12 morbidly obese and 13 non-obese) patients will be enrolled in the study. Morbidly obese and nonobese patients are matched individually 1:1 by age (±10 years), sex, and renal function (as defined by creatinine levels in the urine). There are 4 phases in the clinical study: the pretreatment (screening/baseline) phase of up to 21 days; the 2-day open-label treatment phase when each patients receives a single 2-hour intravenous (directly into the vein) infusion of ceftobiprole 500 mg followed by multiple (up to 15) blood and urine samples drawn over the 24 hours following study drug administration; and the follow-up phase of approximately 1 week after the last blood sample when each patient will be monitored by telephone for development of new adverse events and assessment of ongoing adverse events. Each patient receives a single 2-hour infusion (directly into the vein) of ceftobiprole 500 mg

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) =or > 40 kg/m2 or normal BMI between 18-30
* Blood pressure 90-140 mm
* Non-smoker

Exclusion Criteria:

* History of medically significant illness
* Uncontrolled hypertension
* Uncontrolled high blood cholesterol and triglycerides

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2007-08; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
The pharmacokinetics of ceftobiprole in morbidly obese patients and non-obese patients | up to 30 days (up to 21 days screening plus 2 days open-label treatment phase plus 1-week follow-up).

SECONDARY OUTCOMES:
To assess the pharmacodynamics of ceftobiprole in morbidly obese patients and non-obese patients. | Up to 30 days (up to 21 days screening plus 2 days open label treatment phase plus 1-week follow-up)
To assess safety and tolerability of ceftobiprole in order to support dosing recommendations in the morbidly obese population. | Throughout the study from Day -1 through the post-study follow up

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: Open-Label, Single Dose, Parallel Group Pharmacokinetic Study of Ceftobiprole in Morbidly Obese and Non-Obese Subjects — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=770&filename=CR014185_CSR.pdf